CLINICAL TRIAL: NCT03325114
Title: Safety and Efficacy of Chlorthalidone to Reduce Urinary Calcium Excretion in Adolescents/Yount Adult With Type 1 Diabetes
Brief Title: Safety and Efficacy of Chlorthalidone in Type 1 Diabetes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID restrictions prohibit further study activies
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 66282; 1K23DK114477-01 (NIH)
Record Dates: First submitted 2017-10-20; First posted 2017-10-30 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Type 1 Diabetes Mellitus; Hypercalciuria
Keywords: type 1 diabetes; hypercalciuria
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypercalciuria | interventions — Chlorthalidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Chlorthalidone (Other): Chlorthalidone 12.5-50 mg by mouth daily for 4 weeks
  Interventions: Drug: Chlorthalidone

INTERVENTIONS:
Drug: Chlorthalidone — Chlorthalidone 12.5-5 mg by mouth daily for 4 weeks

SUMMARY:
This open-label study will determine if chlorthalidone is safe and effective for the use of reducing urinary calcium excretion over 4 weeks in subjects with type 1 diabetes

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) is associated with increased urinary calcium loss, which may contribute to the low bone mineral density and increased fracture risk observed in patients with this condition. Chlorthalidone is a thiazide-like diuretic that is commonly used to reduce urinary calcium excretion in other conditions such as idiopathic hypercalciuria. Its safety and efficacy has not been specifically tested in an adolescent type 1 diabetes population.

T1D subjects with hypercalciuria and who meet inclusion/exclusion criteria will be given chlorthalidone daily. Blood and urine tests, blood pressure, and glycemic control will be assessed at weekly study visits for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T1D
* Age 12-21 years
* Tanner Stage 2 or greater pubertal development
* Urine calcium excretion ≥ 4 mg/kg/day
* Able to swallow pills

Exclusion Criteria:

* BMI > 99th percentile for age (<18 years) or BMI >35 kg/m2 (≥ 18 years)
* Coexistent conditions that may affect calcium metabolism including:

  * celiac disease
  * Graves' Disease
  * Addison's disease
  * hypo- or hyperparathyroidism
* History of diabetes related complications including:

  * neuropathy
  * retinopathy
  * nephropathy
  * gastroparesis
* History of oral or inhaled corticosteroid use for ≥ 5 consecutive days within the past month
* History of any diuretic use within the past month
* Laboratory abnormalities on screening bloodwork including:

  * estimated glomerular filtration rate <90 mL/min per 1.73 m2 of body surface area
  * serum calcium >10.5 mg/dL
  * serum potassium <3.5 mmol/L
* Systolic or diastolic blood pressure <5th percentile for age and sex50 for age <18 years or systolic <90 mmHg or diastolic blood pressure <60 mmHG for age ≥18 years

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will be available in aggregate. No plan to share individual data at present.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chlorthalidone
Started | 1
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Due to only one participant being enrolled there are concerns regarding patient confidentiality, therefore no data is being reported.
Arm/Group | Chlorthalidone
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Urinary Calcium Excretion
Description: Change in 24 hour urine calcium excretion
Time Frame: Assessed at baseline and at 4 weeks
Population: as for baseline characteristics
Arm/Group | Chlorthalidone
Number analyzed (Participants) | 0

2. Primary Outcome: Hypokalemia
Description: Serum potassium decreased to <3.5 milliequivalent/L
Time Frame: Assessed weekly for up to 4 weeks or until hypokalemia develops
Population: as for baseline characteristics
Arm/Group | Chlorthalidone
Number analyzed (Participants) | 0

3. Primary Outcome: Hypercalcemia
Description: Serum calcium increased to >10.5 mg/dL
Time Frame: Assessed weekly for up to 4 weeks or until hypercalcemia develops
Population: as for baseline characteristics
Arm/Group | Chlorthalidone
Number analyzed (Participants) | 0

4. Primary Outcome: Hyperglycemia
Description: Change in serum fructosamine
Time Frame: Assessed at baseline and at 4 weeks
Population: as for baseline characteristics
Arm/Group | Chlorthalidone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Due to only one participant being enrolled there are concerns regarding patient confidentiality, therefore no data is being reported.
Arm/Group | Chlorthalidone
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT03325114/Prot_SAP_001.pdf